CLINICAL TRIAL: NCT02316990
Title: China Survey of Stress Ulcer Bleeding in Critically Ill Neurosurgical Patients
Acronym: SUP
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D1843R00056
Record Dates: First submitted 2014-12-11; First posted 2014-12-15 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Stress Ulcers; Stress-related Mucosal Disease (SRMD)
MeSH Terms: conditions — Duodenal Ulcer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients ≥18 ,Neurosurgical departments and whose GCS≤10[4]: The subject population that will be included in the NIS are the consecutive discharged patients ≥18 years old who were hospitalized to Neurosurgical departments and whose GCS≤10[4] within 24 hours of lesion/admission.(GCS: Glasgow Coma Scale NIS: Non-Interventional Study
  )

SUMMARY:
Stress ulcers or stress-related mucosal disease (SRMD) is defined as "acute superficial inflammation lesions of the gastric mucosa induced when an individual is subject to abnormally elevated physiologic demands."[1] Studies have shown that SRMD occurred in 75%-100% ICU patients[1]. Gastrointestinal bleeding due to SRMD is an important complication in critically ill patients. The frequency of clinically important bleeding ranged from 5.3% to 33%.[2] The mortality in ICU patients with stress related bleeding approaches 50%, which is much higher than the patients without bleeding (9%). [3] In 1999, the American Society of Health-System Pharmacists (ASHP) published guidelines on the use of stress ulcer prophylaxis in medical, surgical, respiratory, and pediatric ICU patients [2]. PPIs and H2RA are widely used in China current clinical practice for the prevention of stress ulcer bleeding. However, there is no epidemiology data to show the risk factors for stress ulcer bleeding and the bleeding rate of Chinese neurosurgical critically ill patients who are usually suffering from brain trauma, cerebral haemorrhage or brain tumour operation. Information is needed to know about the characteristics in Chinese critically ill neurosurgical patients.

Objectives of this Non-Interventional Study Primary

1. Primary objective: To estimate the overall incidence of upper gastrointestinal (GI) bleeding in critically ill neurosurgical patients in China.
2. Main secondary objective

   * To estimate the incidence of upper GI bleeding with clinically significant complications in critically ill neurosurgical patients in China.
   * To estimate the incidence of any overt upper GI bleeding without clinically significant complications in critically ill neurosurgical patients in China.
   * To assess time to upper GI bleeding after a cerebral lesion.
   * To investigate potential risk factors associated with upper GI bleeding, and assess how common certain risk factors occurred in upper GI bleeding patients.
   * To assess the overall incidence of upper GI bleeding in critically ill patients by different risk factors for upper GI bleeding.
   * To investigate the drugs, the route of administration, the doses and the duration commonly used for stress ulcer prophylaxis.
   * To investigate the proportion of ICU patients with nasogastric tube, and the duration of nasogastric tube.

(ICU: Intensive care unit PPIs: Proton pump inhibitors H2RA: H2 receptor antagonist)

ELIGIBILITY:
Inclusion Criteria:

* The subject population that will be included in the NIS are the consecutive discharged patients ≥18 years old who were hospitalized to Neurosurgical departments. Those whose Glasgow Coma Scale (GCS) ≤10[4] within 24 hours of lesion/admission will be defined as critically ill patients. Three kinds of cases will be included: brain trauma critically ill patients, cerebral haemorrhage critically ill patients or postoperative brain tumour critically ill patients.

Exclusion Criteria:

* If participating in any clinical trial, the subject cannot take part in this study. Subjects are ineligible if they have below conditions:

  1. Those who were likely to swallow blood (for example, those with severe facial trauma or epistaxis;
  2. Patients with previous total gastrectomy;
  3. Known upper GI lesions that might bleed (e.g., varices, polyps, tumours, etc);
  4. Evidence of active GI bleeding including oesophageal and gastric variceal bleeding, Peptic Ulcer Disease (PUD)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The subject population that will be included in the NIS are the consecutive discharged patients ≥18 years old who were hospitalized to Neurosurgical departments and whose GCS≤10[4] within 24 hours of lesion/admission. The subjects will be focused on brain trauma, cerebral haemorrhage or postoperative brain tumour population.
Sampling Method: Probability Sample
Enrollment: 1416 (Actual)
Dates: Start 2015-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
The primary variable is the overall incidence of upper GI bleeding in critically ill neurosurgical patients | during the first 14 days (up to 14 days) after the cerebral lesion (trauma, haemorrhage or postoperative).

SECONDARY OUTCOMES:
The incidence of upper GI bleeding with clinically significant complications in critically ill neurosurgical patients | during the first 14 days (up to 14 days) after the cerebral lesion (trauma, haemorrhage or postoperative).

CONTACTS AND LOCATIONS:
Locations (11):
- China (11):
  - Research Site, Beijing, Beijing Municipality
  - Research Site, Fuzhou, Fujian
  - Research Site, Tangshan, Hebei
  - Research Site, Changsha, Hunan
  - Research Site, Changchun, Jilin
  - Research Site, Jinan, Shandong
  - Research Site, Shanghai, Shanghai Municipality
  - Research Site, Xi’an, Shanxi
  - Research Site, Chengdu, Sichuan
  - Research Site, Tianjin, Tianjin Municipality
  - Research Site, Hangzhou, Zhejiang

REFERENCES:
- [Derived] Wei J, Jiang R, Li L, Kang D, Gao G, You C, Zhang J, Gao L, Huang Q, Luo D, Zhao G, Zhang H, Wang S, Wang R. Stress-related upper gastrointestinal bleeding in adult neurocritical care patients: a Chinese multicenter, retrospective study. Curr Med Res Opin. 2019 Feb;35(2):181-187. doi: 10.1080/03007995.2018.1448261. Epub 2018 May 30. PMID 29499622
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3094&filename=D1843R00056StudyReportSynopsisV2.0.pdf